CLINICAL TRIAL: NCT03633526
Title: A Phase 3 Study Evaluating the Pharmacokinetics, Safety, and Tolerability of VX-659/TEZ/IVA Triple Combination Therapy in Cystic Fibrosis Subjects 6 Through 11 Years of Age
Brief Title: Evaluation of VX-659/TEZ/IVA in Cystic Fibrosis Subjects 6 Through 11 Years of Age
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study discontinued after Part A due to Sponsor's discretion.
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VX18-659-106; 2018-001711-67 (EudraCT Number)
Record Dates: First submitted 2018-07-27; First posted 2018-08-16 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VX-659/TEZ/IVA (Experimental): Participants who received VX-659 120 milligram (mg)/TEZ 50 mg/ IVA 75 mg as fixed-dose combination (FDC) in the morning and IVA 75 mg as a mono tablet in the evening in the triple combination (TC) treatment period.
  Interventions: Drug: VX-659/TEZ/IVA; Drug: IVA

INTERVENTIONS:
Drug: VX-659/TEZ/IVA — VX-659/TEZ/IVA FDC tablet.
  Other Names: VX-659/VX-661/VX-770; VX-659/tezacaftor/ivacaftor
Drug: IVA — IVA mono tablet.
  Other Names: VX-770; ivacaftor

SUMMARY:
This study will evaluate the pharmacokinetics (PK), safety, tolerability, efficacy, and pharmacodynamic effect of VX-659, tezacaftor (TEZ), and ivacaftor (IVA) when dosed in triple combination (TC) in Cystic Fibrosis (CF) subjects with F/F or F/MF genotypes.

The study was discontinued after completion of Part A due to Sponsor's discretion.

ELIGIBILITY:
Key Inclusion Criteria:

* Homozygous or heterozygous for F508del mutation (F/F or F/MF genotypes)
* Forced expiratory volume in 1 second (FEV1) value ≥40% of predicted mean for age, sex, and height.

Key Exclusion Criteria:

* Clinically significant cirrhosis with or without portal hypertension
* Lung infection with organisms associated with a more rapid decline in pulmonary status.
* Solid organ or hematological transplantation.

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-01-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Children's Hospital Colorado, Aurora, Colorado
  - Ann & Robert Lurie Children's Hospital of Chicago, Chicago, Illinois
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Clinical Research of Charlotte, Charlotte, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 18 participants were enrolled in this study. Two participants were enrolled but were not dosed in triple combination (TC) treatment period. Therefore, results are reported for 16 participants.
Pre-assignment Details: This study was conducted in participants with cystic fibrosis (CF) 6-11 years of age. The study was terminated before start of Part B at Sponsor's discretion.
Groups:
- VX-659/TEZ/IVA: Participants who received VX-659 120 mg/TEZ 50 mg/ IVA 75 mg as FDC in the morning and IVA 75 mg as a mono tablet in the evening for 15 days in the TC treatment period.
Period: Overall Study
Arm/Group | VX-659/TEZ/IVA
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | VX-659/TEZ/IVA
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.2 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax) of VX-659, TEZ, and IVA
Time Frame: Day 1 and Day 15
Population: Pharmacokinetic (PK) set included participants who received at least 1 dose of study drug and for whom the primary PK data were considered to be sufficient and interpretable. Here "Number analyzed" signifies those subjects who were evaluable at the specified timepoint.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | VX-659/TEZ/IVA
Number analyzed (Participants) | 16
microgram per milliliter (mcg/mL)
  VX-659: Day 1: number analyzed (Participants) | 15
  VX-659: Day 1 | 1.81 (0.858)
  VX-659: Day 15: number analyzed (Participants) | 15
  VX-659: Day 15 | 2.55 (1.21)
  TEZ: Day 1: number analyzed (Participants) | 15
  TEZ: Day 1 | 4.53 (1.65)
  TEZ: Day 15: number analyzed (Participants) | 15
  TEZ: Day 15 | 5.22 (1.69)
  IVA: Day 1: number analyzed (Participants) | 15
  IVA: Day 1 | 0.536 (0.208)
  IVA: Day 15: number analyzed (Participants) | 15
  IVA: Day 15 | 0.733 (0.256)

2. Primary Outcome: Observed Pre-Dose Concentration (Ctrough) of VX-659, TEZ, and IVA
Time Frame: Day 8 and Day 15
Population: PK set. Here "Number analyzed" signifies those participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | VX-659/TEZ/IVA
Number analyzed (Participants) | 16
mcg/mL
  VX-659: Day 8 | 0.358 (0.259)
  VX-659: Day 15: number analyzed (Participants) | 15
  VX-659: Day 15 | 0.367 (0.283)
  TEZ: Day 8 | 0.897 (0.488)
  TEZ: Day 15: number analyzed (Participants) | 15
  TEZ: Day 15 | 0.740 (0.421)
  IVA: Day 8 | 0.289 (0.195)
  IVA: Day 15: number analyzed (Participants) | 15
  IVA: Day 15 | 0.283 (0.241)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to 6 Hours (AUC0-6h) of VX-659, TEZ, and IVA
Time Frame: Day 1 and Day 15
Population: PK set. Here "Number analyzed" signifies those participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: hour*mcg/mL (h*mcg/mL)
Arm/Group | VX-659/TEZ/IVA
Number analyzed (Participants) | 16
hour*mcg/mL (h*mcg/mL)
  VX-659: Day 1: number analyzed (Participants) | 15
  VX-659: Day 1 | 5.41 (3.65)
  VX-659: Day 15: number analyzed (Participants) | 15
  VX-659: Day 15 | 8.55 (4.50)
  TEZ: Day 1: number analyzed (Participants) | 15
  TEZ: Day 1 | 15.5 (5.36)
  TEZ: Day 15: number analyzed (Participants) | 15
  TEZ: Day 15 | 19.3 (7.26)
  IVA: Day 1: number analyzed (Participants) | 15
  IVA: Day 1 | 1.64 (0.795)
  IVA: Day 15: number analyzed (Participants) | 15
  IVA: Day 15 | 2.95 (1.18)

4. Secondary Outcome: Maximum Observed Concentration (Cmax) of TEZ Metabolite (M1-TEZ), and IVA Metabolite (M1-IVA)
Time Frame: Day 1 and Day 15
Population: PK set. Here "Number analyzed" signifies those subjects who were evaluable at the specified timepoint.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | VX-659/TEZ/IVA
Number analyzed (Participants) | 16
mcg/mL
  M1-TEZ: Day 1: number analyzed (Participants) | 15
  M1-TEZ: Day 1 | 1.63 (0.553)
  M1-TEZ: Day 15: number analyzed (Participants) | 15
  M1-TEZ: Day 15 | 5.04 (1.27)
  M1-IVA: Day 1: number analyzed (Participants) | 15
  M1-IVA: Day 1 | 1.25 (0.449)
  M1-IVA: Day 15: number analyzed (Participants) | 15
  M1-IVA: Day 15 | 1.73 (0.741)

5. Secondary Outcome: Observed Pre-Dose Concentration (Ctrough) of TEZ Metabolite (M1-TEZ), and IVA Metabolite (M1-IVA)
Time Frame: Day 8 and Day 15
Population: PK set. Here "Number analyzed" signifies those participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | VX-659/TEZ/IVA
Number analyzed (Participants) | 16
mcg/mL
  M1-TEZ: Day 8 | 3.56 (1.33)
  M1-TEZ: Day 15: number analyzed (Participants) | 15
  M1-TEZ: Day 15 | 3.35 (1.23)
  M1-IVA: Day 8 | 0.816 (0.491)
  M1-IVA: Day 15: number analyzed (Participants) | 15
  M1-IVA: Day 15 | 0.858 (0.672)

6. Secondary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to 6 Hours (AUC0-6h) of TEZ Metabolite (M1-TEZ), and IVA Metabolite (M1-IVA)
Time Frame: Day 1 and Day 15
Population: PK set. Here "Number analyzed" signifies those participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: h*mcg/mL
Arm/Group | VX-659/TEZ/IVA
Number analyzed (Participants) | 16
h*mcg/mL
  M1-TEZ: Day 1: number analyzed (Participants) | 15
  M1-TEZ: Day 1 | 5.52 (2.87)
  M1-TEZ: Day 15: number analyzed (Participants) | 15
  M1-TEZ: Day 15 | 25.2 (7.70)
  M1-IVA: Day 1: number analyzed (Participants) | 15
  M1-IVA: Day 1 | 3.60 (1.87)
  M1-IVA: Day 15: number analyzed (Participants) | 15
  M1-IVA: Day 15 | 6.98 (2.94)

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: From first dose of study drug in TC treatment period up to 28 days after last dose of study drug or to the completion of study participation date, whichever occurs first (up to 6 weeks)
Population: Safety set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | VX-659/TEZ/IVA
Number analyzed (Participants) | 16
Participants
  Participants with AEs | 13
  Participants with SAEs | 1

ADVERSE EVENTS:
Time Frame: From first dose of study drug in TC treatment period up to 28 days after last dose of study drug or to the completion of study participation date, whichever occurs first (up to 6 weeks)
Arm/Group | VX-659/TEZ/IVA
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 13/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VX-659/TEZ/IVA (N=16)
Rash (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VX-659/TEZ/IVA (N=16)
Abdominal discomfort (Gastrointestinal disorders) | 1
Post-tussive vomiting (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Chills (General disorders) | 1
Fatigue (General disorders) | 3
Pyrexia (General disorders) | 2
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Procedural anxiety (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 1
Bacterial test positive (Investigations) | 1
Human rhinovirus test positive (Investigations) | 1
International normalised ratio increased (Investigations) | 1
Prothrombin time prolonged (Investigations) | 1
Pulmonary function test decreased (Investigations) | 1
Respirovirus test positive (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Nasal discharge discolouration (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Rash vesicular (Skin and subcutaneous tissue disorders) | 1
Hot flush (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated before start of Part B due to sponsor discretion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT03633526/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/26/NCT03633526/SAP_001.pdf